CLINICAL TRIAL: NCT01565278
Title: Effect of n-3 Polyunsaturated Fatty Acid Lipid Emulsion on Parenteral Nutrition Associated Liver Disease
Brief Title: Fish Oil for Patients With Liver Disease Due to Parenteral Nutrition
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No more eligible patients could be identified.
Sponsor: Johane Allard (Other)
Collaborators: ASPEN Rhoads Research Foundation (Industry); Fresenius Kabi (Industry); University of Alberta (Other); Foothills Medical Centre (Other); St. Boniface Hospital (Other); Hamilton Health Sciences Corporation (Other); St. Paul's Hospital, Canada (Other)
Responsible Party: Sponsor-Investigator, Johane Allard, Professor of Medicine, Gastroenterologist, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-0298-B; 151342 (Other: Health Canada NOL Control Number); 155516 (Other: Health Canada Amendment control #); 161875 (Other: Health Canada Amendment control #); 169378 (Other: Health Canada Amendment control #)
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Total Parenteral Nutrition-induced Cholestasis
Keywords: Parenteral nutrition; fish oil; liver disease; Omegaven; hepatic; liver biopsy; bilirubin
MeSH Terms: conditions — Hyperphagia; Liver Diseases | interventions — Soybean Oil; soybean oil, phospholipid emulsion; Fish Oils; fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soybean oil + Fish oil (Experimental): Intralipid (0.25 g/kg/TPN day) + Omegaven (0.4 g/kg/TPN day) for a period of 6 months.
  Interventions: Drug: Soybean oil + Fish oil
- Soybean oil (Standard treatment) (Active Comparator): Standard treatment: Intralipid (0.25 g/kg/TPN day) for a period of 6 months
  Interventions: Drug: Soybean oil (Standard treatment)

INTERVENTIONS:
Drug: Soybean oil (Standard treatment) — 1. Standard treatment: Soybean oil based emulsion: 0.25 g/kg/TPN day
  Other Names: Intralipid
  Arms: Soybean oil (Standard treatment)
Drug: Soybean oil + Fish oil — Intralipid+Omegaven: 0.25 g/kg/TPN Intralipid day+0.4 g/kg/TPN Omegaven day for 6 months
  Other Names: Intralipid, Omegaven
  Arms: Soybean oil + Fish oil

SUMMARY:
Patients who are not able to eat normally for a longer time require parenteral nutrition, i.e. they receive liquids and nutrients directly into their veins. This can have many long-term side effects, including liver problems. This study will examine whether a specific lipid emulsion containing fish oil can improve liver disease in patients on parenteral nutrition. The investigators will compare changes in bilirubin and liver enzymes after 3 months in 10 patients receiving standard lipid emulsion to 10 patients receiving standard lipids + a fish-oil containing emulsion. The investigators will also assess liver histology, the kind of fat, oxidative stress and gene expression in the liver at the beginning and after 6 months of fish-oil. The investigators also want to compare the baseline values from all 20 patients to 20 healthy controls. This will help to explain how fish oil may improve liver disease in patients on parenteral nutrition.

DETAILED DESCRIPTION:
Chronic exposure to total parenteral nutrition (TPN) can cause parenteral nutrition associated liver disease (PNALD), a progressive condition that may severely affect the liver and lead to end-stage liver disease. Fish oil has been shown to exert beneficial effects as it favorably alters metabolism and inflammation. It has been used parenterally (Omegaven) in young children with short bowel syndrome and PNALD with encouraging results. In adults it has mostly been used in peri-surgical settings as well as in critically ill patients, again proving its effectiveness.

The goal of this proposal is to show that Omegaven use in home-TPN patients with PNALD and elevated bilirubin despite conventional treatment, is beneficial in improving cholestasis and reducing intrahepatic inflammation. Primary objective is to compare the response to treatment between the Omegaven and the Intralipid group. Secondary objectives are to study the effect of Omegaven supplementation on single liver function tests, liver histology, liver fatty acid composition, liver oxidative stress and gene expression. In addition, the investigators want to compare the baseline values of all 20 patients to 20 healthy controls subjects.

After establishing that the patients' liver disease does not improve with conventional medical treatments for 3 months, as evidenced by repeated blood work at that time, they will all have a liver biopsy done as per diagnostic standards. They will then be randomized to either continue receiving Intralipid (0.25 g/kg/TPN day) or a mixture of Intralipid (0.25 g/kg/TPN day) and Omegaven (0.4 g/kg/TPN day) for a period of 3 months. After that, patients in the Omegaven arm will continue their treatment for 3 more months. Those in the Intralipid arm will be switched over to also receive Omegaven for the following 6 months.

Blood work will be repeated every 3 months after the initiation of the intervention. A repeat liver biopsy will be done in both groups after 6 months.

Main outcome is response to treatment (improvement in liver function tests) after 3 months (comparing Intralipid to Omegaven). In addition, change in liver function tests during the 6 months on Omegaven will be assessed. Lipid peroxidation and oxidative stress, fatty acid composition, and gene expression in the liver will be compared before and after 6 months on Omegaven.

In a second part of the study baseline values from all 20 patients will be compared to 20 healthy controls. Controls will be recruited from the healthy living liver donor transplant program at the University Health Network (UHN). Liver samples will be obtained at the time of hepatectomy for transplantation. The same measurements as for the patient livers will be performed in healthy liver tissue.

Significance: The investigators aim to reveal the beneficial effects of fish oil supplementation in the setting of PNALD. Should this pilot study show improvement in the liver disease with Omegaven, a larger, randomized trial should follow. Comparison with healthy controls will provide further insight into the pathogenesis of PNALD, which to date is not completely understood

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable patients on home TPN with PNALD with persistently elevated bilirubin (>1.5 times > normal) for at least 3 months despite standard treatment with ursodeoxycholic acid (15-30 mg/kg or at least 500 mg/d orally), changes in TPN (reduction to 25 kcal/kg/TPN day with Intralipid 0.25 g/kg) , and antibiotics (Metronidazole 500 mg bid and Ciprofloxacin 500 mg bid)
* male or female,equal or over 18 years of age
* on stable TPN regimen equal or over 3 days/week
* on a stable drug regimen for equal or over 3 months prior to randomization, which will not changed for the study duration if these drugs are ursodeoxycholic acid given for PNALD or others affecting glucose and lipid metabolism

Exclusion Criteria:

* Not receiving lipid emulsion as part of TPN
* Allergy to fish, egg , soy, and peanuts
* Liver disease of other etiology (e.g. excessive alcohol intake >20g/d, viral hepatitis, auto-immune or drug-induced, hemochromatosis, alfa 1-antitrypsin deficiency, Wilson's disease)
* Complications of chronic liver disease, such as recurrent variceal bleeding, ascites, encephalopathy or any other reason contraindicating a liver biopsy
* Severe hemorrhagic disorders
* Sepsis - Inflammatory processes
* Taking medications that precipitate steatohepatitis (e.g. corticosteroids, methotrexate, or amiodarone)
* Pregnancy, lactation
* Fluid restriction - Omegaven is more dilute than Intralipid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Response to treatment at 3 months | 3 months
  Response is defined as improvement of at least one PNALD parameter by 20% or more; PNALD parameters are: ALP, GGT, ALT, total bilirubin Yes/No

SECONDARY OUTCOMES:
Change in total and conjugated bilirubin over time | 0, 3, 6 months on Omegaven
Changes in liver function test (ALP, AST, GGT) over 6 months | 0, 3, 6 months on Omegaven
Changes in liver histology between baseline and 6 months on Omegaven | 0, 6 months on Omegaven
Changes in liver fatty acid composition between baseline and 6 months on Omegaven | 0, 6 months on Omegaven
  Fatty acid composition by gas chromatography
Changes in liver oxidative stress between baseline and 6 months | 0, 6 months
  Lipid peroxides in liver tissue (test-kit)
Changes in hepatic gene expression between baseline and 6 months on Omegaven | 0, 6 months on Omegaven
  Hepatic gene expression (mRNA) by microarray

OTHER OUTCOMES:
Insulin resistance | 0, 3, 6, 9 months
  HOMA-insulin resistance 0, 3, 6 months in Omegaven group 0, 3, 6, 9 months in Intralipid-group switching to Omegaven after 3 months
Blood lipid profile | 0, 3, 6, 9 months
  Triglycerides, total cholesterol, LDL, HDL 0, 3, 6 months in Omegaven group 0, 3, 6, 9 months in Intralipid-group switching to Omegaven after 3 months
Complete blood count (CBC) | 0, 3, 6, 9 months
  0, 3, 6 months in Omegaven group 0, 3, 6, 9 months in Intralipid-group switching to Omegaven after 3 months
international normalized ratio (INR) | 0, 3, 6, 9 months
  0, 3, 6 months in Omegaven group 0, 3, 6, 9 months in Intralipid-group switching to Omegaven

CONTACTS AND LOCATIONS:
Overall Officials: Johane P Allard, MD,FRCPC, Principal Investigator — University Health Network, Toronto
Locations (4):
- Canada (4):
  - Foothills Medical Center, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - St Boniface Hospital, Winnipeg, Manitoba
  - University Health Network, Toronto, Ontario

REFERENCES:
- [Background] Raman M, Gramlich L, Whittaker S, Allard JP. Canadian home total parenteral nutrition registry: preliminary data on the patient population. Can J Gastroenterol. 2007 Oct;21(10):643-8. doi: 10.1155/2007/217897. PMID 17948134
- [Background] Fernandes G, Kaila B, Jeejeebhoy KN, Gramlich L, Armstrong D, Allard JP. Canadian home parenteral nutrition (HPN) registry: validation and patient outcomes. JPEN J Parenter Enteral Nutr. 2012 Jul;36(4):407-14. doi: 10.1177/0148607111434599. Epub 2012 Feb 10. PMID 22326909
- [Background] Jurewitsch B, Gardiner G, Naccarato M, Jeejeebhoy KN. Omega-3-enriched lipid emulsion for liver salvage in parenteral nutrition-induced cholestasis in the adult patient. JPEN J Parenter Enteral Nutr. 2011 May;35(3):386-90. doi: 10.1177/0148607110382023. PMID 21527601
- [Background] Kelly DA. Intestinal failure-associated liver disease: what do we know today? Gastroenterology. 2006 Feb;130(2 Suppl 1):S70-7. doi: 10.1053/j.gastro.2005.10.066. PMID 16473076
- [Background] Guglielmi FW, Boggio-Bertinet D, Federico A, Forte GB, Guglielmi A, Loguercio C, Mazzuoli S, Merli M, Palmo A, Panella C, Pironi L, Francavilla A. Total parenteral nutrition-related gastroenterological complications. Dig Liver Dis. 2006 Sep;38(9):623-42. doi: 10.1016/j.dld.2006.04.002. Epub 2006 Jun 12. PMID 16766237
- [Background] Messing B, Joly F. Guidelines for management of home parenteral support in adult chronic intestinal failure patients. Gastroenterology. 2006 Feb;130(2 Suppl 1):S43-51. doi: 10.1053/j.gastro.2005.09.064. PMID 16473071
- [Background] Diamond IR, Sterescu A, Pencharz PB, Kim JH, Wales PW. Changing the paradigm: omegaven for the treatment of liver failure in pediatric short bowel syndrome. J Pediatr Gastroenterol Nutr. 2009 Feb;48(2):209-15. doi: 10.1097/MPG.0b013e318182c8f6. PMID 19179884
- [Background] Calhoun AW, Sullivan JE. Omegaven for the treatment of parenteral nutrition associated liver disease: a case study. J Ky Med Assoc. 2009 Feb;107(2):55-7. PMID 19263944
- [Background] Chung PH, Wong KK, Wong RM, Tsoi NS, Chan KL, Tam PK. Clinical experience in managing pediatric patients with ultra-short bowel syndrome using omega-3 fatty acid. Eur J Pediatr Surg. 2010 Mar;20(2):139-42. doi: 10.1055/s-0029-1238283. Epub 2010 Feb 22. PMID 20178080
- [Background] Fallon EM, Le HD, Puder M. Prevention of parenteral nutrition-associated liver disease: role of omega-3 fish oil. Curr Opin Organ Transplant. 2010 Jun;15(3):334-40. doi: 10.1097/mot.0b013e3283394879. PMID 20503524